CLINICAL TRIAL: NCT04478409
Title: Characterization of a Functional Test for Mediterranean Family Fever Screening - 2
Acronym: DEPIST-FMF 2
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0236
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Familial Mediterranean Fever; MEFV Gene Mutation
Keywords: Familial Mediterranean fever; Interleukin-1β; MEFV gene mutation; innate immunity
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sample will be code and sent to the laboratory within 24 hours (Inserm U1111, Lyon). For healthy subjects, research does not involve drawing additional blood from their blood donation.
  There will be no long-term storage or establishment of biological collections. The monocytes will be extracted, selected and counted. The pyras inflammasome will then be activated and the interleukin-1β secretion will be measured by ELISA. Cell death will be quantified in real time by fluorimetry.
  Validation on cellular models in vitro: immortalized monocytes will be invalidated for the MEFV gene by CrispR-Cas9 and different inducible variants of the MEFV gene will be expressed in MEFV knot out cells. These genetically modified cells will then undergo the tests for stimulation of the inflammatory Pyrine according to the same procedures as the monocytes of the patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children or adult with Familial Mediterranean fever: Considering 5 clearly pathogenic (homozygous) genotypes, 15 possibly pathogenic genotypes (5 pathogenic mutations in the heterozygous state, 10 possibly pathogenic mutations in the homozygous or heterozygous state), a number of 80 patients will be necessary to cover the correlation analysis genotype / phenotype.
  The study does not change the usual course of care. Only an additional blood sample (4 ml for children under 12 and 10 ml for children 12 and over and adults) during a planned blood test is specific to research (no risk added). The benefit / risk balance therefore remains unchanged with regard to the usual care of patients.
  Interventions: Biological: one additional blood sample during a planned blood test
- Healthy blood donor: Healthy blood donor

INTERVENTIONS:
Biological: one additional blood sample during a planned blood test — The study does not change the usual course of care. Only an additional blood sample (4 ml for children under 12 and 10 ml for children 12 and over and adults) during a planned blood test is specific to research (no risk added). The benefit / risk balance therefore remains unchanged with regard to the usual care of patients.
  Groups: Children or adult with Familial Mediterranean fever

SUMMARY:
Familial Mediterranean fever (FMF) is the most common auto-inflammatory disease (prevalence: 1-5 / 10,000 inhabitants). It is caused by mutations in the MEFV gene, which encodes variants of the Pyrine inflammasome. Inflammasomes are protein complexes of the innate immunity that produce pro-inflammatory cytokines (interleukin-1β).

In vitro, our preliminary results demonstrated that the activation of the inflammatory pyrine (measured by the concentration of interleukin-1β) by kinase inhibitors is significantly increased in FMF patients compared to healthy subjects. Furthermore, a measurement of cell death gave significant results in differentiating the patients from the controls.

The performance of this functional has been tested, fast and simple diagnostic test on common mutations and wish to assess its characteristics for MEFV mutations.

The investigators hypothesize that this quick and simple functional test can serve as a diagnostic tool for FMF and can quantitatively discriminate against patients with different mutations (genotypes).

ELIGIBILITY:
Inclusion Criteria:

* Children 4 years of age or older or adults
* Having a clinical picture compatible with an FMF and a previous genetic analysis finding at least one mutation of the MEFV gene pathogenic or possibly pathogenic for the FMF group;
* Newly diagnosed or in the process of follow-up (with no time limit or evolutionary criteria);
* During specific or non-specific treatment of the disease or without treatment;
* For whom a blood test is planned as part of routine care;
* Whose informed non-opposition has been collected (or parental non-opposition in the case of a minor patient);

Exclusion Criteria:

* Person under legal protection or under the protection of justice or any other protective measures;
* Person out of state to express their consent;
* Person in emergency situation, vital or not;
* Known infections with HIV and / or HBV and / or HCV;

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will involve 80 patients with Familial Mediterranean fever, presenting a previous genetic analysis finding at least one mutation of the MEFV gene, considered pathogenic or possibly pathogenic (60 heterozygotes or complex mutations and 20 homozygotes). The controls will be 80 healthy subjects (French national medical and scientific center (INSERM) and French blood bank (EFS) convention).
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Quantification of interleukin-1β | At inclusion
  quantification of the capacity of the concentration of interleukin-1β measured in the supernatants of primary monocytes in response to kinase inhibitors, to discriminate between FMF subjects among themselves according to genotypes, and among control subjects (healthy subjects).
  All samples will be analysed in the INSERM Unit 1111 - CIRI Centre International de Recherche en Infectiologie - Lyon - Team Inflammasome, bacterial infections and autoinflammation.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Hôpital Femme-Mère-Enfant, Bron
  - CH de Versailles - Hôpital André Mignot, Le Chesnay
  - Hôpital Edouard Herriot, Lyon
  - Hôpital de la Croix-Rousse, Lyon
  - CHU de Montpellier, Montpellier
  - Service de Pédiatrie - CHU de Nîmes - Hôpital Carémeau, Nîmes
  - Hôpital Tenon, Paris
  - Hôpital Lyon Sud, Pierre-Bénite